CLINICAL TRIAL: NCT00004363
Title: Study of the Pathogenesis and Pathophysiology of Familial Neurohypophyseal Diabetes Insipidus
Status: Completed | Type: Observational
Sponsor: National Center for Research Resources (NCRR) (NIH)
Collaborators: Northwestern University (Other)
Other Study IDs: NCRR-M01RR00048-0568; NU-568
Record Dates: First submitted 1999-10-18; First posted 1999-10-19 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2003-12

CONDITIONS: Diabetes Insipidus; Diabetes Insipidus, Neurohypophyseal
Keywords: diabetes insipidus; endocrine disorders; rare disease
MeSH Terms: conditions — Diabetes Insipidus; Diabetes Insipidus, Neurogenic; Endocrine System Diseases; Rare Diseases | interventions — Chlorpropamide; Deamino Arginine Vasopressin

INTERVENTIONS:
Drug: chlorpropamide
Drug: desmopressin

SUMMARY:
OBJECTIVES: I. Determine whether diverse mutations of the vasopressin-neurophysin II (AVP-NPII) gene cause autosomal dominant familial neurohypophyseal diabetes insipidus by directing the production of an abnormal preprohormone.

II. Determine whether the AVP-NPII gene-directed preprohormone accumulates and destroys magnocellular neurons because it cannot be folded and processed efficiently.

DETAILED DESCRIPTION:
PROTOCOL OUTLINE: This project involves 2 clinical studies. Members of known kindreds participate in Study I; members of kindreds who have not been surveyed, genotyped, or phenotyped participate in Study II.

In Study I, participants undergo clinical, hormonal, radiologic, and biochemical studies. Assessment on unrestricted fluid intake includes body weight, urine volume, osmolality, creatinine, sodium, potassium, urea, glucose, arginine-vasopressin (AVP), oxytocin, and aquaporin-II.

Participants with diabetes insipidus (DI) undergo a standard fluid deprivation test; those without DI undergo standard water load and hypertonic saline testing.

Previously untreated DI patients may be given intranasal or subcutaneous desmopressin or oral chlorpropamide (adults only) for 2 or 3 days.

Magnetic resonance imaging of the pituitary-hypothalamic area is performed on all patients with and without gadolinium.

Infants and children are studied annually for the first 5 years or until they develop DI. Affected adults are studied every 2-5 years. Unaffected adults are re-tested only if they subsequently report de novo symptoms suggestive of DI.

In Study II, participants undergo similar genotype and phenotype testing. Kindreds demonstrating the familial neurohypophyseal diabetes insipidus phenotype and genotype are added to Study I. Kindreds found to have a different type of DI are directed into a companion protocol.

ELIGIBILITY:
* Verified or suspected familial neurohypophyseal diabetes insipidus with or without an identified mutation of the vasopressin-neurophysin II gene Affected and unaffected members of kindreds entered

Ages: 6 Months to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1995-12

CONTACTS AND LOCATIONS:
Overall Officials: Gary L. Robertson, Study Chair — Northwestern University
Locations (1):
- Northwestern University Medical School, Chicago, Illinois, United States

REFERENCES:
- [Background] Hansen LK, Rittig S, Robertson GL. Genetic basis of familial neurohypophyseal diabetes insipidus. Trends Endocrinol Metab. 1997 Nov;8(9):363-72. doi: 10.1016/s1043-2760(97)00157-4. PMID 18406826
- [Background] Rittig S, Robertson GL, Siggaard C, Kovacs L, Gregersen N, Nyborg J, Pedersen EB. Identification of 13 new mutations in the vasopressin-neurophysin II gene in 17 kindreds with familial autosomal dominant neurohypophyseal diabetes insipidus. Am J Hum Genet. 1996 Jan;58(1):107-17. PMID 8554046
- [Background] McLeod JF, Kovacs L, Gaskill MB, Rittig S, Bradley GS, Robertson GL. Familial neurohypophyseal diabetes insipidus associated with a signal peptide mutation. J Clin Endocrinol Metab. 1993 Sep;77(3):599A-599G. doi: 10.1210/jcem.77.3.8370682.